CLINICAL TRIAL: NCT03853616
Title: A Phase I Safety, Dose Finding and Feasibility Trial of MB-CART19.1 in Patients With Relapsed or Refractory CD19 Positive B Cell Malignancies
Brief Title: MB-CART19.1 r/r CD19+ B-cell Malignancies (BCM)
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Miltenyi Biomedicine GmbH (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M-2017-322; 2017-002848-32 (EudraCT Number)
Record Dates: First submitted 2019-02-19; First posted 2019-02-25 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Lymphoblastic Leukemia Recurrent; B-cell Lymphoma Recurrent; B-cell Lymphoma Refractory; Chronic Lymphocytic Leukemia Recurrent; Chronic Lymphocytic Leukemia Refractory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- DL 0: 1x10e5 MB-CART19.1 cells (Experimental): In each dose level of each of the three cohorts three 3 + 3 patients will be treated. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD.
  Interventions: Biological: MB-CART19.1
- DL 1: 5x10e5 MB-CART19.1 cells (Experimental): Dose evaluation will start in Cohorts 1 and 2 with Dose Level 1. In each dose level of each of the three cohorts three 3 + 3 patients will be treated. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD.
  Interventions: Biological: MB-CART19.1
- DL 2: 1x10e6 MB-CART19.1 cells (Experimental): Dose evaluation will start in Cohort 3 with Dose Level 2, sparing Dose Level 1. If Dose Level 2 is not tolerated, Dose Level 1 will be tested. In each dose level of each of the three cohorts three 3 + 3 patients will be treated. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD.
  Interventions: Biological: MB-CART19.1
- DL 3: 3x10e6 MB-CART19.1 cells (Experimental): In each dose level of each of the three cohorts three 3 + 3 patients will be treated. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD. In Dose Level 3, three additional patients will be treated, if no DLT occurred. Dose Level 0 will be tested only if Dose Level 1 is not tolerable.
  Interventions: Biological: MB-CART19.1

INTERVENTIONS:
Biological: MB-CART19.1 — MB-CART19.1 consists of autologous CD19 Chimeric Antigen Receptor (CAR) transduced CD4/CD8 enriched T cells targeting CD19-positive tumor cells in b cell malignancies
  Other Names: CD19-targeting CAR T cells; Anti-CD19 CAR T cells

SUMMARY:
This is a phase l multi-centric, single arm, prospective open, dose-escalation study in patients with relapsed or refractory CD19-positive B cell malignancies (ALL, NHL, CLL). The trial will include adult and pediatric patients. In total approximately 48 patients will be included in the trial. There will be three individual cohorts, defined by disease biology: pediatric ALL and aggressive pediatric NHL (Cohort 1), adult ALL (Cohort 2) and adult NHL/CLL (Cohort 3).

DETAILED DESCRIPTION:
This trial will evaluate the safety of the MB-CART19.1 and determine the recommended dose levels for each of the three disease cohorts.

Dose evaluation will start in Cohorts 1 and 2 with Dose Level 1 and in Cohort 3 with Dose Level 2, sparing Dose Level 1 (see figure 1). Each of the cohorts will evaluate the safety of MB-CART19.1.

In each dose level of each of the three cohorts three 3 + 3 patients will be treated. A particular dose level will be expanded to 6 patients if one patient out of 3 patients treated at that particular dose level develops DLT. Once this occurs, further dose-escalations are halted until the dose has proven to be safe in the expanded cohort. If 2 or more in a cohort of 6 patients develop DLT no further dose escalation is allowed, and the next lower dose level will be expanded to 6 patients in total. The highest dose among the dose levels tested at which no more than one out of six patients experiences DLT will be considered the MTD. In Dose Level 3, three additional patients will be treated, if no DLT occurred. Dose Level 0 will be tested only if Dose Level 1 is not tolerable.

Cohort 3 will Start with Dose Level 2. If Dose Level 2 is not tolerated, Dose Level 1 will be tested. DLT will be evaluated within 4 weeks after the infusion of MB-CART19.1. An interval of at least 28 days between the treatment of the first and the second patient in each dose level (and in each cohort) is mandatory.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients must have r/r CD19-expressing ALL or NHL/CLL
* CD19 expression must be detected on the malignant cells by flow cytometry (leukemia, malignant effusion in NHL) or immunohistochemistry (NHL);
* Age ≥ 1 year (if deemed fit by treating investigator);
* Absolute CD3+ T cell count ≥100/μl;
* ECOG performance score of 0-2 if >16 years old, or Lansky performance score of >50 if ≤16 years old at screening;
* No active Hepatitis B, Hepatitis C, HIV1/2;
* No childbearing potential or negative pregnancy test at screening and before chemotherapy in women with childbearing potential;
* Signed and dated informed consent/assent by patients
* and meet the following disease-specific criteria:

ALL:

* patients with >5% blasts in BM (M2 or M3) after at least one standard chemotherapy and one salvage regimen who are ineligible for allogeneic stem cell transplant (alloSCT) or have refractory disease activity precluding alloSCT at this time, or
* patients who have relapsed post alloSCT at least 100 days posttransplant, with no evidence of active GVHD, and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
* patients with Ph+ ALL if they are intolerant to tyrosine kinase inhibitor (TKI) therapy, or if they have r/r disease after treatment with at least 2 different TKIs.
* ALL patients with combined bone marrow and CNS and/or testicular relapse are eligible only if the extramedullary disease has been successfully cleared by conventional therapy at the time of inclusion (e.g. intrathecal chemotherapy, orchiectomy).

Pediatric aggressive NHL (1-17 years):

* patients after at least one salvage chemotherapy as bridge to alloSCT or
* patients ineligible for alloSCT or
* patients who have relapsed post alloSCT at least 100 days posttransplant, with not evidence of active GVHD, and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
* patients with CNS disease (excluding isolated CNS lymphoma) are eligible only if disease has been successfully cleared by intrathecal chemotherapy at the time of inclusion.

Adult NHL:

* patients after at least one standard chemotherapy and one salvage regimen as bridge to alloSCT or
* patients who are ineligible for alloSCT or
* patients who have relapsed post alloSCT at least 100 days posttransplant, with no evidence of active GVHD, and no longer taking immunosuppressive agents for at least 30 days prior to enrollment.
* patients with CNS disease (excluding isolated CNS lymphoma) are eligible only if disease has been successfully cleared by intrathecal chemotherapy at the time of inclusion.

CLL:

* patients with r/r disease after established and approved treatment options have failed.
* patients not eligible or appropriate for conventional alloSCT.

Exclusion Criteria:

* Isolated CNS or testicular relapse in ALL;
* Isolated CNS lymphomas;
* Active solid brain metastases or history of solid brain metastases
* Current autoimmune disease, or history of autoimmune disease with potential CNS involvement;
* Active clinically significant CNS dysfunction (including but not limited to uncontrolled seizure disorders, cerebrovascular ischemia or hemorrhage, dementia, paralysis);
* History of an additional malignancy other than non-melanoma skin cancer or carcinoma in situ unless disease free for ≥3 years;
* Pulmonary function: Patients with pre-existing severe lung disease or an oxygen requirement of >28% O2 supplementation or active pulmonary infiltrates on chest X-ray;
* Cardiac function: Fractional shortening <28% or left ventricular ejection fraction <50% by echocardiography;
* Renal function: GFR ≤29 mL/min/1.73 m2 by CKD-EPI for patients 18 yrs (Levey et al. 2009) or creatinine clearance ≤29 mL/min/1.73 m2 by Schwartz formula (Schwartz et al. 1976) for patients <18 yrs of age;
* Liver function: Patients with a serum bilirubin >3 times upper limit of normal or an AST or ALT > 5 times upper limit of normal, unless due to leukemic liver infiltration in the estimation of the investigator;
* Rapidly progressive disease that in the estimation of the investigator would compromise ability to complete study therapy;
* Pregnant or breast-feeding females;
* Medications:

  * Systemic chemotherapies, corticosteroids with the exception of physiologic replacement dosing, tyrosine kinase inhibitors (TKI) within 7 days prior to leukapheresis,
  * Fludarabine/clofarabine or immunosuppressive drugs and antibodies (e.g. rituximab, calcineurin inhibitors, blinatumomab) or investigational drugs or donor lymphocyte transfusions or radiation therapy within 30 days prior to apheresis,
  * Alemtuzumab within 3 months prior to leukapheresis,
  * Exception: Intrathecal chemotherapy is allowed prior to treatment, but should be discontinued in ALL and BL 10 days prior to MB-CART19.1 infusion to limit risk of neurotoxicities;
* Hypersensitivity against any drug or its ingredients/impurities that is scheduled or likely to be given during trial participation, e.g. as part of the mandatory lymphodepletion protocol, pre-medication for infusion, rescue medication/salvage therapies for treatment related toxicities;
* Intake of concomitant medication contraindicated for other reasons than hypersensitivity, e.g. live vaccines and fludarabine;
* Contraindication of trial related procedures as judged by the investigator, e.g. lumbar punctures for CSF sampling;
* Female patients of child-bearing potential not willing to practice a highly effective form of birth control from the time of enrollment and for 12 months after dosing the IMP;
* Male patients of fathering potential not willing to practice a highly effective form of birth control from the time of enrollment and for 12 months after dosing the IMP;
* Concurrent participation in another interventional trial that could interact with this trial, e.g. CAR T trials;
* Cerebral dysfunction, legal incapacity of adult patients;
* Committal to an institution on judicial or official order.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Determination of the recommended dose of MB-CART19.1 | until day 28 after infusion of MB-CART19.1
  Maximum tolerated dose (MTD), defined as the highest dose level of the two to three dose levels tested at which <33% of patients experience DLT until day 28 after infusion of MB-CART19.1, on the basis of safety and toxicity assessment of MB-CART19.1 per adverse events (AE) reporting classified according to CTCAE version 5.0.

SECONDARY OUTCOMES:
Overall incidence and severity of adverse events | through study completion, an average of 5 years
  per adverse events (AE) reporting classified according to CTCAE version 5.0
Response to treatment for each timepoint | day 28
  ORR in ALL (Rate of CR/CRh)
Response to treatment for each timepoint | day 28, week 12, month 6, 1 year
  Rate MRD-negative CR in ALL
Response to treatment for each timepoint | day 28, patients not in CR on day 28: month 3
  ORR in NHL/CLL (Rate of CR/PR)
Occurence of B-cell depletion | through study completion, an average of 5 years
  Circulating B cell numbers
Phenotype and persistence of MB-CART19.1 | days 2, 7, 10, 14, 28, weeks 8, 12, months 6, 12, 24, 36, 48, 60
  Blood samples for determination of persistence/phenotyping of infused MB-CART19.1 will be analysed
Number of patients with successful MB-CART19.1 production | day 0
  Number of patients meeting the inclusion criteria and none of the exclusion criteria for who an autologous MB-CART19.1 product can be generated
Rate of ALL patients achieving MRD negative CR | day 28, week 12, month 6, 1 year
  Rate MRD-negative CR in ALL
Duration of response | through study completion, an average of 5 years
  Determination of response rate
Disease-free survival | at 1 year after MB-CART19.1 infusion in patients not receiving alloSCT
  disease-free survival at 1 year after adoptive immunotherapy with MB-CART19.1 in patients not receiving alloSCT
Overall survival | at 1 year after MB-CART19.1 infusion in patients not receiving alloSCT
  overall survival at 1 year after adoptive immunotherapy with MB-CART19.1 in patients not receiving alloSCT

CONTACTS AND LOCATIONS:
Overall Officials: Claudia Rössig, Prof. Dr., Principal Investigator — Univeristy Hospital Muenster
Locations (9):
- Germany (9):
  - Charité - University clinic, pediatric clinic with focus on oncology and hematology, Berlin
  - Universitätsklinikum Erlangen, Erlangen
  - University medicine Goettingen, Clinic of hematology and medical oncology, Göttingen
  - Children's Hospital of Dr. von Hauner by Ludwig-Maximilian University, Munich
  - Universitätsklinikum Münster - Klink für Kinderheilkunde und Jugendmedizin / Pädiatrische Hämatologie und Onkologie, Münster
  - Universitätsklinikum Münster - Medizinische Klinik A / KMT Zentrum, Münster
  - Tuebingen University clinic, medical university clinic for internal medicine, Tübingen
  - University clinic for children and youth medicine, Tübingen
  - University clinic, pediatric hematology and oncology, Würzburg

IPD SHARING:
Plan to Share IPD: No